CLINICAL TRIAL: NCT04146285
Title: A Phase I Clinical Trial of BAT4406F Injection on the Safety, Tolerability, and Pharmacokinetics in Patients With Neuromyelitis Optica Spectrum Disorders
Brief Title: A Phase I Clinical Trial of BAT4406F Injection in Patients With Neuromyelitis Optica Spectrum Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT-4406F-001-CR
Record Dates: First submitted 2019-09-26; First posted 2019-10-31 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2023-03

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BAT4406F (Experimental)
  Interventions: Drug: BAT4406F

INTERVENTIONS:
Drug: BAT4406F — Open-label dose escalation starting from 20mg.
  Route of administration: intravenous infusion.

SUMMARY:
This study is a phase I clinical study of the safety, tolerability, and pharmacokinetics of BAT4406F injection in patients with neuromyelitis optica spectrum disorders.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, dose-escalation study in NMOSD patients in which subjects will receive BAT4406F injection via intravenous infusion. A 3 + 3 design will be utilized to define a maximum tolerated dose (MTD). The overall objective is to assess the safety, tolerability, and pharmacokinetics of BAT4406F injection in NMOSD patients.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with the NMOSD diagnostic criteria developed by the 2015 International NMO Diagnostic Team (IPND);
* 18-65 years old , male or female;
* At least 2 relapses occurred within 2 years before screening, or at least 1 relapse within 1 year before screening;
* Discontinue the immunosuppressive agents such as azathioprine within 28 days before the baseline;
* EDSS score ≤ 6;
* Men and women with fertility must agree to use effective methods of contraception during treatment and within 12 months of treatment completion;
* Agree to participate in the trial and sign the informed consent in writing.

Exclusion Criteria:

* Any monoclonal antibody treatment was used within 6 months prior to dosing;
* Having been treated with anti-CD20 monoclonal antibody;
* Live vaccine received within 4 weeks before screening;
* Having participated in another clinical study within 1 month or 5 half-lives of the drug prior to the baseline (whichever is longer);
* A history of allergies to monoclonal antibodies; severe allergic reaction to certain foods or drugs;
* Abnormal liver function, kidney function and bone marrow reserve;
* HIV-positive history or HIV-positive at screening; hepatitis B and/or hepatitis C history or hepatitis B surface antigen-positive at screening; or hepatitis C virus (HCV) antibody positive; treponema pallidum antibody positive when enrolled;
* History of infections that investigators have identified as unsuitable for testing;
* Patients with a clear history of heart disease ;
* Have a history of mental disorders;
* Pregnant or lactating women, and female subjects who have a positive pregnancy test at screening;
* None of the investigators or their relatives participating in the study could be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity（DLT） | 4weeks
  Safety and tolerability endpoint
Maximum tolerated dosed (MTD) | up to 6 months
  Safety and tolerability endpoint
Area under the curve (AUC) | up to 6 months
  Pharmacokinetic endpoint
Maximum serum drug concentration (Cmax) | up to 6 months
  Pharmacokinetic endpoint
Half-life period(t1/2) | up to 6 months
  Pharmacokinetic endpoint
Maximum serum drug time (Tmax) | up to 6 months
  Pharmacokinetic endpoint
CD19+ B lymphocyte ratio | up to 6 months
  Pharmacodynamics endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Xiangjun Chen, Principal Investigator — Huashan Hospital; Jing Zhang, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yu H, Chen Y, Qi Y, Yang H, Cao G, Yang W, Li S, Yang X, Wang H, Zhang J, Chen X. First-in-Human Study of BAT4406F, an ADCC-Enhanced Fully Humanized Anti-CD20 Monoclonal Antibody in Patients With Neuromyelitis Optica Spectrum Disorders. CNS Neurosci Ther. 2024 Nov;30(11):e70126. doi: 10.1111/cns.70126. PMID 39592888